CLINICAL TRIAL: NCT04242173
Title: A Single Arm Phase II Study of Cemiplimab-rwlc in Immunocompromised Patients With Unresectable Locally Recurrent and/or Metastatic Cutaneous Squamous Cell Carcinoma (CSCC)
Brief Title: Cemiplimab-rwlc for Unresectable Locally Recurrent and/or Metastatic CSCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Interest
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20114
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Cutaneous Squamous Cell Carcinoma of the Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cemiplimab-rwlc treatment (Experimental): Immunocompromised patients will be given Cemiplimab-rwlc every 3 weeks
  Interventions: Drug: Cemiplimab-Rwlc

INTERVENTIONS:
Drug: Cemiplimab-Rwlc — Cemiplimab-rwlc will be administered as a flat dose of 350 mg IV over approximately 30 minutes every 21 days (+/- 3 days)
  Other Names: Libtayo

SUMMARY:
The purpose of this research study is to determine how people with weakened immune systems and unresectable (cannot be removed by surgery) locally recurrent and/or metastatic cutaneous squamous cell carcinoma (CSCC) respond to study treatment with Cemiplimab. Cemiplimab is approved for sale in United States by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive Cutaneous Squamous Cell Carcinoma (CSCC)
* Immunocompromised patients with invasive CSCC. Immunocompromised patients are defined as: (a) History of HIV with CD4 counts >/= 200 and no AIDS-defining illness (b) History of treated or active hematologic malignancies including lymphoma, Hodgkin's disease, chronic lymphocytic leukemia, chronic myeloid leukemia, multiple myeloma, and myeloproliferative neoplasm.
* At least 1 lesion that is measurable by study criteria by RECIST 1.1. Externally visible cutaneous Squamous Cell Cancer (SCC) target lesion(s) greater than >10 mm, bi-dimensional measurements of the external lesion(s) with a color photograph may be used as target lesions.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Laboratory values as defined per protocol
* Ability to sign informed consent
* Ability and willingness to comply with scheduled visits, treatment plans, laboratory tests, and other study-related procedures.
* CSCC not amenable to surgery or radiation therapy such as unresectable tumors determined by surgeons, surgical morbidity unacceptable by the patients, inability to deliver radiation safely determined by radiation oncologists, or radiation related toxicities unacceptable by the patients.

Note: In lieu of individual consults performed during screening, it will suffice to document the contraindication of surgery and radiation therapy via a clinic note from the investigator indicating that an individualized benefit:risk assessment was performed by a multidisciplinary team (consisting of, at minimum, a radiation oncologist AND EITHER a medical oncologist with expertise in cutaneous malignancies OR a dermato-oncologist, OR a head and neck surgeon) within 60 days prior to enrollment in the proposed study, and the radiation therapy was deemed to be contraindicated. This is not required for patients with distant metastatic disease.

Exclusion Criteria:

* Prior known allergy to Cemiplimab-rwlc
* Prior exposure to PD-1 or PD-L1 inhibitors
* Prior exposure to idelalisib
* Immunocompromised patients due to solid organ transplant, allogenic bone marrow transplant, and/or autoimmune disease.
* Untreated brain metastasis(es) that may be considered active.
* Immunosuppresive corticosteroid doses (>10 mg prednisone daily or equivalent for >5 consecutive days) within 4 weeks prior to the first dose of Cemiplimab-rwlc.
* Known active infection requiring therapy, including acute infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). However, it is not required to test only to determine the eligibility for the trail. As an exception, known HIV infection is allowed.
* History of pneumonitis within the last 5 years.
* Grade >/= 3 hypercalcemia at time of enrollment
* Patients on any systemic anticancer treatment (chemotherapy, targeted systemic therapy, photodynamic therapy), investigational or standard of care for CSCC within 28 days of the initial administration of Cemiplimab-rwlc are excluded.
* Patients on any systemic anticancer treatment (chemotherapy, targeted systemic therapy, photodynamic therapy), investigational or standard of care for non-hematologic malignancy within 28 days of the initial administration of Cemiplimab-rwlc or planned to occur during the study period are excluded.

NOTE: (a) Patients receiving bisphosphonates or denosumab are not excluded. (b) Patients receiving maintenance or supportive therapies for their hematological malignancies are not excluded. (c) If the patients have been disease free for >2 years, patients receiving adjuvant hormonal therapies for breast cancer, prostate cancer, or thyroid cancer are not excluded.

* Patients who cannot discontinue the concurrent use of other chemopreventive agents such as 5-FU, capecitabine, Efudex, imiquimod, acitretin are not allowed.
* Radiation therapy within 7 days of initial administration of Cemiplimab-rwlc or planned to occur during the study period.
* Breast feeding
* Positive serum pregnancy test (a false positive pregnancy test, if demonstrated by serial measurements and negative ultrasound, will not be exclusionary)
* Concurrent non-hematologic malignancy other than cutaneous SCC within 3 years of date of first planned dose of Cemiplimab-rwlc , except for tumors with negligible risk of metastasis or death, such as adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast, or low-risk early stage prostate adenocarcinoma (T1-T2a N0 M0 and Gleason score ≤6 and PSA ≤10 ng/mL) for which the management plan is active surveillance, or prostate adenocarcinoma with biochemical-only recurrence with documented PSA doubling time of > 12 months for which the management plan is active surveillance.
* Any acute or chronic psychiatric problems that, in the opinion of the investigator, make the patient ineligible for participation.
* Continued sexual activity in men or women of childbearing potential who are unwilling to practice highly effective contraception during the study and until 6 months after the last dose of study drug. Note: Highly effective contraceptive measures include stable use of oral contraceptives such as combined estrogen and progestogen and progestogen only hormonal contraception or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal ligation; vasectomy, and sexual abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine H Chung, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cemiplimab-rwlc Treatment
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early due to lack of interest
Arm/Group | Cemiplimab-rwlc Treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) as indicated by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 analysis of radiologic scans. In some patients, response assessments include photos and radiologic scans and will be evaluated by composite efficacy criteria.
  Clinical lesions will only be considered measurable when they are superficial (eg, skin nodules and palpable lymph nodes) and ≥10 mm (≥1 cm) diameter as assessed using calipers (e.g., skin nodules). Patients who are deemed as not evaluable according to RECIST 1.1 or inevaluable by the composite efficacy criteria will be considered as not reaching ORR.
Time Frame: Up to 12 months
Population: Data was not collected due to low number of patients accrued to study
Arm/Group | Cemiplimab-rwlc Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS), defined as time from on study date to disease progression
Time Frame: Up to 12 months
Population: Data was not collected due to low number of patients accrued to study
Arm/Group | Cemiplimab-rwlc Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS), defined as time from on study date to death from any cause
Time Frame: Up to 12 months
Population: Data was not collected due to low number of patients accrued to study
Arm/Group | Cemiplimab-rwlc Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment to 30 days after end of treatment, approximately 7 months
Arm/Group | Cemiplimab-rwlc Treatment
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cemiplimab-rwlc Treatment (N=3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT04242173/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04242173/ICF_001.pdf